CLINICAL TRIAL: NCT03930329
Title: Mindfulness-based Treatment to Prevent Smoking Relapse: a Pilot Randomized Controlled Study
Brief Title: Mindfulness-based Treatment to Prevent Smoking Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tung Wah Group for Hospital Integrated Centre (Unknown)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NTEC-2019-smoke
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRP group (Experimental): The mindfulness-based relapse prevention program consists of eight weekly 2-hour sessions. It combines mindfulness with evidence-based cognitive behavioural techniques that help participants to recognize internal and external triggers of their substance abuse, including smoking. Each session consists of mindful practices with cognitive exercises. The standardized treatment manual was published
  Interventions: Behavioral: MBRP group
- usual care (No Intervention): All participants in this trial will receive usual care, which consists of 8-12 weeks of counselling and drug treatment to help smokers quit. Data from the centre shows that approximately 50% of smokers are successfully abstinent from smoking at end of the program, as confirmed by the carbon monoxide breath test. This trial will only recruit those who successfully quitted smoking. During this 8-12 week program, written information about relapse prevention is given, including information for maintaining healthy lifestyles (e.g. diet/sleep/exercise/emotional control). Participants will receive follow-up phone interviews by trained smoking cessation counsellors at end of the program (week 8-12)

INTERVENTIONS:
Behavioral: MBRP group — same as arm description
  Arms: MBRP group

SUMMARY:
Background: Smoking causes a variety of health problems and causes burden to healthcare systems. Even when support is provided, local data suggest that around 50% of biochemically confirmed quitters resume smoking within 6 months of participating in a smoking cessation program. Mindfulness-based intervention is a promising option because accumulating evidence from randomized controlled trials support its use among smokers. Our team aims to determine if mindfulness-based interventions can prevent relapse in smokers who recently quit smoking. A pilot trial is needed to determine the feasibility of recruitment, randomisation and acceptability of the intervention in these patients Method: Forty participants, who just quitted smoking, will be randomised in a 1:1 ratio to the 8week mindfulness-based relapse prevention (MBRP) program and to usual care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* self-reported smokers
* can speak and read Cantonese and Chinese
* willing to participate in at least 7 of the 8 sessions of the MBRP program

Exclusion Criteria:

* pregnancy (they will have different motivations for quitting smoking)
* significant physical illness or severe cognitive impairment that prevents communication, such as blindness or severe hearing loss, because mindfulness exercise instructions are given verbally and reading materials are given out after each class
* history of psychotic disorders or symptoms, because MBRP is not confirmed safe or effective in this group of patients
* suicidal tendency as detected by PHQ-9 (see below)
* we will not exclude participants with mood disorders for the reasons stated in the introduction, but participants with drug changes for their mood disorders in the last 3 months will be excluded (ethics approval and informed consent will be obtained for assessing patients' medical records, CMS of the hospital authority or e-health, to confirm drug information)
* active illicit drug use and
* past mindfulness course or practices in the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
the rate of retention | recruitment and thoughout the 8-week program
  As a pilot study to test the feasibility of the future RCT, the primary outcomes will include the rates of recruitment and retention. The amount of homework completed will be self-reported using a homework diary
rate of recruitment | from recruitment to the start of the 8-week program
  As a pilot study to test the feasibility of the future RCT, the primary outcomes will include the rates of recruitment and retention.

SECONDARY OUTCOMES:
reported abstinence from smoking during the last seven days, which will be confirmed with an expired carbon monoxide level of <6 ppm | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  reported abstinence from smoking during the last seven days, which will be confirmed with an expired carbon monoxide level of <6 ppm
9-item Patient Health Questionnaire (PHQ-9) | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument for depressive symptoms
7-item Generalized Anxiety Disorder Questionnaire (GAD-7) | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument for anxiety symptoms
the Alcohol Use Identification Test (AUDIT) | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument for alcohol use
10-item Perceived Stress Scale | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument for stress level; there are two factors: (i) perceived helplessness and (ii) perceived efficacy; each subscales' score can be calculated by adding up scored from individual questions; Perceived helplessness subscale score: 0-24 (higher is worse); perceived efficacy subscale score 0-16 (higher the better) total score calculation: reverse scoring for questions in 'self-efficacy' sub-scale, total score can be calculated by adding all the scores together; Theoretical rage: 0 to 40; The higher the score, the higher the perceived stress
20-item Positive Affect and Negative Affect Scale | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument for positive and negative affect; 10 item for positive items and 10 for negative items; score range from 10-50 for both items. For total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect
Minnesota Nicotine Withdrawal Scale | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  no subscale; total score is the sum of the score of individual item; possible score: 0-36; the higher the score, the more severe the withdrawal symptoms
Five-Facet Mindfulness Questionnaire (FFMQ) | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  validated instrument to assess the level of mindfulness; 5 subscale; each subscale score is calucated by adding score from individual items; the protocol had included reverse scoring for item 3, 5, 8, 10, 12, 13, 14, 16, 17, 18, 22, 23, 25, 28, 30, 34, 35, 38, 39. Subscale score: observing (8-40), describe (8-40), act with awareness (8-40), nonjudge (8-40), nonreact (7-35); the higher the score, the higher the degree of mindfulness in each subscale
Brief questionnaire of smoking urges | assessed at baseline (before class 1) and immediately after the eighth MBRP class
  subscale 1 - intention/desire to smoke; subscale 2 - relief of negative affect & urgent desire to smoke; the score of each subscale is calculated by adding the score from individual items; possible scores for each subscale = 5-35; the higher the score, the higher the smoking urge

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Wah Group of Hospitals, Integrated Centre on Smoking Cessation, Tuen Mun Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
will make available on request of investigators